CLINICAL TRIAL: NCT05635955
Title: Remimazolam Versus Propofol, in Combination With Esketamine for Painless Abortion
Brief Title: Remimazolam Versus Propofol for Painless Abortion
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Maternal and Child Health Hospital of Hubei Province (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Li Na, Deputy Chief Physician, Maternal and Child Health Hospital of Hubei Province
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MCHH_001
Record Dates: First submitted 2022-11-15; First posted 2022-12-02 (Actual); Last update posted 2022-12-02 (Actual); Status verified 2022-11

CONDITIONS: Anesthesia; Abortion Early
MeSH Terms: interventions — remimazolam; Propofol; Esketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Remimazolam (Experimental): Intravenous Remimazolam will be co-administrated with esketamine.
  Interventions: Drug: Remimazolam; Drug: Esketamine
- Propofol (Active Comparator): Intravenous Propofol will be co-administrated with esketamine.
  Interventions: Drug: Propofol; Drug: Esketamine

INTERVENTIONS:
Drug: Remimazolam — Total intravenous anaesthesia will be induced with 0.3mg/kg remimazolam and 0.3mg/kg esketamine, slow injection.
  During the painless abortion surgery, if the MOAA/S scores > 1 or body movements occur, supplemental 0.2 mg/kg remimazolam (IV) will be administrated.
  Arms: Remimazolam
Drug: Propofol — Total intravenous anaesthesia will be induced with 2mg/kg propofol and 0.3mg/kg esketamine, slow injection.
  During the painless abortion surgery, if the MOAA/S scores > 1 or body movements occur, supplemental 0.25 mg/kg propofol (IV) will be administrated.
  Arms: Propofol
Drug: Esketamine — 0.3mg/kg esketamine will be co-administrated in both arms

SUMMARY:
The goal of this clinical trial is to compare the efficacy and safety of propofol vs. remimazolam in combine use of esketamine in women with early pregnancy undergoing painless abortion. The main questions it aims to answer are:

* whether remimazolam plus esketamine (R+E) has a better sedative and analgesic effectiveness than propofol plus esketamine (P+E).
* whether R+E has less adverse events than P+E.

Participants will be randomly allocated to two groups: R+E and P+E group.

* For those in group R+E: they will be administered with 0.3mg/kg remimazolam and 0.3mg/kg esketamine before the abortion surgery.
* For those in group P+E: they will be administered with 2mg/kg propofol and 0.3mg/kg esketamine before the abortion surgery.

We will compare R+E with P+E to see if the time to loss of conscious and time to recover from the sedation will be shorter and if there will be less severe adverse events in R+E.

ELIGIBILITY:
Inclusion Criteria:

* early intrauterine pregnancy less than 12 weeks confirmed by transabdominal ultrasound and blood HCG
* the American Society of Anesthesiologists (ASA) physical status ranked I-II
* competent to provide informed consent

Exclusion Criteria:

* chronic pain
* psychiatric disorders
* liver or kidney failure
* severe metabolic disorders
* poor respiratory functions
* cardiovascular diseases

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Time to loss of consciousness | 5 - 30 minutes
  The time from the study drug administration to loss of consciousness

SECONDARY OUTCOMES:
Success rate of sedation | Intraoperative period, 30 minutes - 1.5 hours
  Defined as completing the induction of anesthesia without an additional dosage
Recovery time | Postoperative 30 minutes
  Time to fully awake, defined as by a modified Aldrete score which will be recorded every 3 minutes from the end of the procedure with a recovery index (MAS) of 9 or more.
Mean arterial pressure (MAP) | Intraoperative period, 30 minutes - 1.5 hours
  MAP level will be monitored and recorded at 4 time points, including the entry into the operation room (Time 0), in sedation when vaginal dilator is placed (Time 1), in sedation when curettage begins (Time 2), and postoperative awakening (Time 3).
Heart rate (HR) | Intraoperative period, 30 minutes - 1.5 hours
  HR will be monitored and recorded at 4 time points, including the entry into the operation room (Time 0), in sedation when vaginal dilator is placed (Time 1), in sedation when curettage begins (Time 2), and postoperative awakening (Time 3).
Adverse events | Intraoperative and post-operation, 30 minutes - 1.5 hours
  The adverse events will be monitored and recorded during the operation and post-operation. AE will include: respiratory depression (defined as SpO2< 95%), hypotension (defined as systolic arterial pressure < 80 mmHg, or decreased baseline systolic blood pressure > 20%), hypertension, bradycardia (defined as decrease in HR < 50/min), number of body movements, injection site pain and nausea and vomiting.
Post-operative pain | Post-operation after fully awake, 30 minutes - 1 hour
  It will be assessed by Visual Analogue Scale (VAS) pain score. The VAS consists of a 10cm line, with two end points representing 0 ('no pain') and 10 ('pain as bad as it could possibly be').

CONTACTS AND LOCATIONS:
Overall Officials: Na Li, MD, Principal Investigator — Maternal and Child Health Hospital of Hubei Province
Locations (1):
- Maternal and Child Health Hospital of Hubei Province, Wuhan, Hubei, China